CLINICAL TRIAL: NCT00228930
Title: A Pilot Trial Correlating Metabolic Profile of Tamoxifen With Pharmacogenetic Predictors and Clinical Effects
Brief Title: Tamoxifen Pharmacogenetics and Clinical Effects
Status: Completed | Type: Observational
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Collaborators: Indiana University School of Medicine (Other)
Other Study IDs: 0208-14; U01GM061373-05 (NIH)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Tamoxifen; Prevention
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood Serum Plasma

INTERVENTIONS:
Drug: Tamoxifen (pharmacodynamic analysis) — Tamoxifen 20mg po daily

SUMMARY:
The purpose of this research is to try to identify which women who take tamoxifen are likely to suffer from hot flashes or are more likely to have other side effects or benefits from the drug. The researchers will do so by determining whether there are mutations that normally occur in human DNA that might influence the way individuals respond to medications.

DETAILED DESCRIPTION:
The study will test the following hypotheses.

1. There is a relationship between genetically distinct metabolic profiles of tamoxifen and the frequency and severity of hot flashes in women on chronic tamoxifen therapy.
2. Genetically distinct metabolic profiles for tamoxifen effect lipid profile, bone turnover metabolites and bone mineral density, and coagulation factors.
3. Different genetic profiles of estrogen responsive genes influence the pharmacodynamic effects of tamoxifen in cardiovascular system.

ELIGIBILITY:
Inclusion Criteria:

1. 18-years or older
2. Women with a prior breast cancer or who are at a high risk for developing the disease and about to start tamoxifen therapy.
3. Participants must not be treated with concomitant chemotherapy or hormone therapy other than tamoxifen. They must not have ovarian ablation or currently being treated with radiation therapy and/or chronic corticosteroids.
4. The participant must not be taking anti-hot flash therapy (clonidine, bellergal, megestrol acetate). Vitamin E, selective serotonin reuptake inhibitors, or herbal remedies are allowed provided that the participant has been taking the remedy for at least 4 weeks and intends to continue the remedy for at least the first month while on the study, and allows for one-month follow up evaluation (hot flash diaries and blood samples).
5. The participant must not be pregnant or lactating.
6. The participant is able and willing to sign an informed consent.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients included women 18 years or older, non-pregnant or lactating, who were recommended tamoxifen for adjuvant treatment or for the prevention of breast cancer from the oncology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2002-09; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Flockhart, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - UMCCC, Ann Arbor, Michigan

REFERENCES:
- [Result] Rae JM, Goetz MP, Hayes DF, Ingle JN, Li L, Storniolo AM, Stearns V, Flockhart DA. CYP2D6 genotype and tamoxifen response. Breast Cancer Res. 2005 Jul 29;7(5):E6. doi: 10.1186/bcr1297. No abstract available. PMID 16168100
- [Result] Lim YC, Desta Z, Flockhart DA, Skaar TC. Endoxifen (4-hydroxy-N-desmethyl-tamoxifen) has anti-estrogenic effects in breast cancer cells with potency similar to 4-hydroxy-tamoxifen. Cancer Chemother Pharmacol. 2005 May;55(5):471-8. doi: 10.1007/s00280-004-0926-7. Epub 2005 Feb 1. PMID 15685451
- [Result] Jin Y, Desta Z, Stearns V, Ward B, Ho H, Lee KH, Skaar T, Storniolo AM, Li L, Araba A, Blanchard R, Nguyen A, Ullmer L, Hayden J, Lemler S, Weinshilboum RM, Rae JM, Hayes DF, Flockhart DA. CYP2D6 genotype, antidepressant use, and tamoxifen metabolism during adjuvant breast cancer treatment. J Natl Cancer Inst. 2005 Jan 5;97(1):30-9. doi: 10.1093/jnci/dji005. PMID 15632378
- [Result] Stearns V, Johnson MD, Rae JM, Morocho A, Novielli A, Bhargava P, Hayes DF, Desta Z, Flockhart DA. Active tamoxifen metabolite plasma concentrations after coadministration of tamoxifen and the selective serotonin reuptake inhibitor paroxetine. J Natl Cancer Inst. 2003 Dec 3;95(23):1758-64. doi: 10.1093/jnci/djg108. PMID 14652237
- [Result] Lee KH, Ward BA, Desta Z, Flockhart DA, Jones DR. Quantification of tamoxifen and three metabolites in plasma by high-performance liquid chromatography with fluorescence detection: application to a clinical trial. J Chromatogr B Analyt Technol Biomed Life Sci. 2003 Jul 5;791(1-2):245-53. doi: 10.1016/s1570-0232(03)00218-6. PMID 12798184
- [Derived] Hayes DF, Skaar TC, Rae JM, Henry NL, Nguyen AT, Stearns V, Li L, Philips S, Desta Z, Flockhart DA; Consortium on Breast Cancer Pharmacogenomics (COBRA). Estrogen receptor genotypes, menopausal status, and the effects of tamoxifen on lipid levels: revised and updated results. Clin Pharmacol Ther. 2010 Nov;88(5):626-9. doi: 10.1038/clpt.2010.143. Epub 2010 Sep 8. PMID 20827267
- [Derived] Henry NL, Rae JM, Li L, Azzouz F, Skaar TC, Desta Z, Sikora MJ, Philips S, Nguyen AT, Storniolo AM, Hayes DF, Flockhart DA, Stearns V; Consortium on Breast Cancer Pharmacogenomics Investigators. Association between CYP2D6 genotype and tamoxifen-induced hot flashes in a prospective cohort. Breast Cancer Res Treat. 2009 Oct;117(3):571-5. doi: 10.1007/s10549-009-0309-1. Epub 2009 Jan 20. PMID 19153830
- [Derived] Ntukidem NI, Nguyen AT, Stearns V, Rehman M, Schott A, Skaar T, Jin Y, Blanche P, Li L, Lemler S, Hayden J, Krauss RM, Desta Z, Flockhart DA, Hayes DF; Consortium on Breast Cancer Pharmacogenomics. Estrogen receptor genotypes, menopausal status, and the lipid effects of tamoxifen. Clin Pharmacol Ther. 2008 May;83(5):702-10. doi: 10.1038/sj.clpt.6100343. Epub 2007 Aug 22. PMID 17713466
- See also: The Pharmacogenetics and Pharmacogenomics Knowledge Base — http://www.pharmgkb.org